CLINICAL TRIAL: NCT01655511
Title: A Phase 1, Randomized, Double-Blind, Crossover, Ascending Dose-Tolerance Study To Assess The Safety And Pharmacokinetics Of Tafamidis Doses Greater Than 120 Mg As Oral Solution In Healthy Volunteers
Brief Title: Safety And Pharmacokinetic Assessment Of Orally Administered Tafamidis In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: B3461040; B3461040
Record Dates: First submitted 2012-07-12; First posted 2012-08-02 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: TTR Cardiomyopathy
Keywords: Pharmacokinetic; pharmacodynamic
MeSH Terms: interventions — tafamidis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Period 1 (Experimental): 240 mg tafamidis arm
  Interventions: Drug: Tafamidis
- Period 2 (Experimental): 480 mg arm
  Interventions: Drug: Tafamidis
- Period 3 (Experimental): TBD dose
  Interventions: Drug: Tafamidis

INTERVENTIONS:
Drug: Tafamidis — 240 mg, solution, single dose
  Arms: Period 1
Drug: Tafamidis — 480 mg, solution, single dose
  Arms: Period 2
Drug: Tafamidis — TBD dose will be a single dose if < 720 mg or a loading dose followed by additional dose if > 720 mg.
  Arms: Period 3

SUMMARY:
This study in healthy male and female volunteers will investigate the safety and tolerability of three increasing oral doses of tafamidis

ELIGIBILITY:
Inclusion Criteria:

* Healthy, males or females, 21 to 55 years old.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2.

Exclusion Criteria:

Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).

Condition affecting drug absorption. Blood pressure or ECG abnormalities. Recent treatment with an investigational, prescription, or non-prescription drug

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2012-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of orally administered tafamidis in healthy volunteers at escalating doses >120 mg. Safety assessments will include spontaneous reporting of adverse events, concomitant medications, physical examination, | Day 0 and Day 6
vital signs, ECGs, and clinical laboratory tests. | Day 0 and Day 6

SECONDARY OUTCOMES:
Cmax - Maximum Observed Plasma Concentration (Cmax) | 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, and 120 hrs
tmax - Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, and 120 hrs
AUC0-24 - AreArea under the Concentration-Time Curve (AUC) | 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, and 120 hrs
AUClast - Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)] | 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, and 120 hrs
AUCinf - Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] | 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, and 120 hrs
t½ - Plasma Decay Half-Life (t1/2) | 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, and 120 hrs
Transthyretin blood concentration in mg/dL | Days 0,1,2,3,4,5,6
Transthyretin stabilization (%) | Days 0,1,2,3,4,5,6

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3461040&StudyName=Safety%20And%20Pharmacokinetic%20Assessment%20Of%20Orally%20Administered%20Tafamidis%20In%20Healthy%20Volunteers